CLINICAL TRIAL: NCT03824340
Title: Intracytoplasmic Sperm Injection Preparation in Infertile Women With Unexplained Infertility
Brief Title: Intracytoplasmic Sperm Injection Preparation in Infertile Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aljazeera Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ICSI preparation
Record Dates: First submitted 2019-01-25; First posted 2019-01-31 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Doxycycline

STUDY DESIGN:
Intervention Model Description: A randomized controlled study
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Doxycycline before ICSI (Active Comparator): extra medications (Doxycycline ) group before ICSI : in which Women who will receive the Doxyxycline before ICSI Intervention : Women will receive Doxycycline before ICSI
  Interventions: Drug: Doxycycline before ICSI
- control group (No Intervention): control group : No intervention : in which Women willnot receive the extra medications (Doxycycline ) before ICSI

INTERVENTIONS:
Drug: Doxycycline before ICSI — Extra medication (Doxycycline ) group before ICSI :,women who will receive more medications (Doxycycline ) before starting the ICSI process
  Other Names: Medical treatment with Doxycycline
  Arms: Doxycycline before ICSI

SUMMARY:
Infertility is a common gynecological problem is women

DETAILED DESCRIPTION:
Intracytoplasmic sperm injection is one of the aisted reproduction techniques that help to solve this problem

ELIGIBILITY:
Inclusion Criteria:

* Women who have infertility with age between 20 -42 years

Exclusion Criteria:

* women who has ovarian or endometrial factor of infertility

Ages: 20 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — infertile women
Enrollment: 500 (Estimated)
Dates: Start 2019-01-30 (Actual); Primary Completion 2019-11-30 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
the number of women who will have successful ICSI | within 4 months
  The number of women who will get pregnant after ICSI with extra treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, PhD, Principal Investigator — Algazeerah hospital -Location (Giza -Egypt ) and National Research centre egypt
Locations (1):
- Algazeerah, Giza, Egypt